CLINICAL TRIAL: NCT05210998
Title: Investigation of the Effects of Respiratory Muscle Training Combined With Aerobic Exercise in Persons With Obstructive Sleep Apnea Syndrome
Brief Title: Respiratory Muscle Training Combined With Aerobic Exercise in Obstructive Sleep Apnea Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Seker Abanoz, PhD student, Physioterapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Obstructive Sleep Apnea
Record Dates: First submitted 2021-12-04; First posted 2022-01-27 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-06

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: Sleep Apnea , Respiratory Muscle Training, Aerobic Exercise
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grup 1: (Active Comparator): Combined Exercise Group:
  Gradual aerobic exercise training AND Respiratory muscle training
  Interventions: Other: Gradual Aerobic exercise training AND Respiratory muscle training
- grup 2: (Active Comparator): Aerobic Exercise Group:
  Gradual Aerobic exercise training
  Interventions: Other: Gradual Aerobic exercise training

INTERVENTIONS:
Other: Gradual Aerobic exercise training AND Respiratory muscle training — Combined Exercise Group
  Arms: grup 1:
Other: Gradual Aerobic exercise training — Aerobic exercise Group
  Arms: grup 2:

SUMMARY:
In this study, which was planned to evaluate the effects of inspiratory and expiratory respiratory muscle training in addition to aerobic exercise in individuals with OSAS; 40 cases over the age of 40 who were diagnosed with severe (AHI: 30 and over) Obstructive Sleep Apnea Syndrome by polysomnography in the Sleep Laboratory of the Department of Chest Diseases of the Istanbul University Istanbul Medical Faculty Hospital will be included. The cases will be divided into two groups with the randomization system and the education of both groups will continue for a total of 8 weeks. In the literature, it is stated that there is a need for studies on the benefits and results of the use of respiratory muscle training as an adjunct therapy to CPAP or oral devices. No studies were found that evaluated the effects of inspiratory and expiratory respiratory muscle training in addition to aerobic exercise in patients with OSAS. For this reason, OSAS patients using regular CPAP were planned as two groups in the treatment part of this study. Control Group: For gradual aerobic exercise training, bicycle ergometer training in the hospital environment and brisk walking at home once a week (3 days a week, 20-40 minutes a day) will be given under supervision two days a week.

Training Group: In addition to the aerobic exercise, the training group will be given respiratory muscle training once a day, 5 days a week, as a home program. Intraoral pressure measurements will be repeated once a week to calculate the new threshold load. Respiratory muscle training: Respiratory muscle training in 50% of MIP and 30% of MEP, as ICE + IME (5 days a week, 15 minutes per day, 15 minutes of IMI). Evaluations will be repeated before and after treatment. The original value of this study is that the effects of Respiratory Muscle Training Combined with Aerobic Exercise in addition to CPAP treatment will be investigated in individuals with OSAS.

DETAILED DESCRIPTION:
Combined Exercises Grup: In addition to the aerobic exercise, the training group will be given respiratory muscle training once a day, 5 days a week, as a home program. Intraoral pressure measurements will be repeated once a week to calculate the new threshold load. Respiratory muscle training: Respiratory muscle training in 50% of MIP and 30% of MEP, as ICE + IME (5 days a week, 15 minutes per day, 15 minutes of IMI). Evaluations will be repeated before and after treatment. The original value of this study is that the effects of Respiratory Muscle Training Combined with Aerobic Exercise in addition to CPAP treatment will be investigated in individuals with OSAS.

Aerobic Exercises Grup: For gradual aerobic exercise training, bicycle ergometer training in the hospital environment and brisk walking at home once a week (3 days a week, 20-40 minutes a day) will be given under supervision two days a week Obstructive Sleep Apnea Syndrome (OSAS) is a syndrome with a highly complex pathophysiology characterized by repetitive complete or partial upper airway occlusions during sleep. As a result of collapse in the pharyngeal airways during sleep, air flow to the lungs decreases partially (hypopnea) or completely (apnea), hypoxia and hypercapnia develop, and the congestion ends with the end of sleep. The repetition of these situations that develop during sleep stimulates the sympathetic nervous system and causes changes in blood pressure.Excessive daytime sleepiness and neurocognitive disorders can be observed as a result of sleep disruptions and hypoxia that develop with multiple stimuli .It has been reported that there is a continuous increase in the prevalence of OSAS. The incidence of OSAS in the general adult population varies between 9-38%, with a higher incidence in males. Due to obesity, its prevalence is increasing at an alarming rate, especially in middle and high-income countries . OSAS causes potentially serious health consequences such as impaired quality of life, emotional impairment, neurocognitive impairment, permanent brain damage, cardiovascular morbidity, and sudden death during sleep. OSAS has a very complex pathophysiology and the roles of influencing factors are also variable among individuals. In the physiopathology of upper airway obstruction, factors such as anatomical and mechanical factors, impaired contractile function of upper airway muscles, respiratory control instability come to the fore . One of the mechanisms that cause altered neuromechanical responses in OSAS is the deterioration of the contractile function of the upper airway muscles. In these patients, the upper respiratory tract muscles work under hypoxic conditions and as a result, a modification in the muscle fiber structure develops. In this modification, muscle fibers change from type I fibers that are resistant to fatigue to type II muscle fibers that increase strength but are not resistant to fatigue. As a result, the contractility of the muscle is preserved, but the fatigue increases. With this modification in the muscle fiber, inflammation may occur in the muscle working under increased load, with muscle damage that impairs the contractility of the muscle. Muscle dysfunction may develop as a result of these events .

During sleep, there is a decrease in lung volume and upper airway dilator muscle tone. Therefore, upper and lower airway muscle function is relatively reduced during sleep and may increase airway obstruction. It is thought that increasing upper airway dilator muscle activity and increasing lung volume are effective in maintaining airway patency. Coordinated contraction of the upper airway dilator muscles (eg genioglossus) and inspiratory pump muscles (eg diaphragm) is required for breathing to continue with an open airway. Inspiratory muscle weakness increases susceptibility to hypoventilation during sleep .

Treatment methods of OSAS include conservative (Continuous Positive Airway Pressure (CPAP) device and intraoral device applications) and surgical interventions. CPAP therapy, which is the most effective method available in OSAS, has been shown to improve sleepiness, hypertension and many cardiovascular indices seen in patients . CPAP is considered the first choice in the treatment of especially moderate or severe OSAS cases, but it is costly and patient compliance is an important condition that affects treatment success.

It is known that respiratory muscle training increases respiratory muscle strength in people with COPD and neuromuscular diseases . It has been reported that inspiratory muscle training in OSAS patients improves OSAS severity, daytime sleepiness and sleep quality, decreases the severity and frequency of snoring, improves respiratory muscle strength, and can reduce the cost of CPAP treatment by increasing its use in rehabilitation programs. However, it has been shown that training applied to the upper respiratory tract with the didgeridoo instrument in people with snoring and OSAS reduces daytime sleepiness, apnea-hypopnea index, and upper airway collapse. Strengthening both inspiratory and expiratory muscles seems reasonable given that weakness of the upper airway and inspiratory muscles in these patients affects sleep-related outcome measures. In addition, it is stated in the literature that there is a need for studies on the benefits and results of the use of respiratory muscle training as an adjunct to CPAP or oral devices .

It is known that most of the patients with OSAS also have low exercise capacity. OSAS severity is associated with worsening exercise tolerance. In the treatment of OSAS patients, exercise training in addition to CPAP therapy has received increasing attention in recent years . It has been shown that regular exercise training applied in patients with OSAS reduces AHI, body weight and body mass index, improves aerobic capacity and quality of life . In a recent meta-analysis, aerobic exercise training has been reported to effectively improve quality of life, daytime sleepiness, and sleep quality . No studies were found that evaluated the effects of inspiratory and expiratory respiratory muscle training in addition to aerobic exercise in patients with OSAS. The aim of this study is to evaluate the effects of inspiratory and expiratory respiratory muscle training in addition to aerobic exercise in patients with OSAS.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with Severe Obstructive Sleep Apnea
2. Being over 40 years old
3. Using CPAP
4. Not to be included in any exercise and diet program throughout the study

Exclusion Criteria:

1. Unstable angina pectoris,
2. Body Mass Index (BMI)>35 kg/m2
3. Chronic Lung Disease
4. Neurological or musculoskeletal problems that prevent him from exercising
5. Psychiatric disorder (eg, Bipolar disorder, schizophrenia)
6. Unstable cardiovascular conditions
7. Unstable metabolic conditions

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Polysomnography (PSG) | 8 weeks
  Polysomnography is the gold standard diagnostic test for the diagnosis of adult patients with suspected OSAS based on a comprehensive sleep assessment. It is also used to evaluate the severity of OSAS and the effectiveness of treatment.Patients over the age of 40, who were diagnosed with severe (AHI: 30 and above) Obstructive Sleep Apnea Syndrome by a Chest Diseases Specialist by polysomnography in the Sleep Laboratory of the Chest Diseases Department of the Istanbul University Istanbul Medical Faculty Hospital, will be included in the study. Polysomnography is routinely performed in the Sleep Laboratory in the diagnosis and follow-up of patients with OSAS.

SECONDARY OUTCOMES:
Respiratory Muscle Strength Assessment. | 8 weeks
  In the evaluation of respiratory muscle strength, mouth pressure measurement method will be used in accordance with ATS/ERS criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Medical Faculty, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Eckert DJ, Malhotra A, Jordan AS. Mechanisms of apnea. Prog Cardiovasc Dis. 2009 Jan-Feb;51(4):313-23. doi: 10.1016/j.pcad.2008.02.003. PMID 19110133
- [Background] Hsia JC. Anatomy and physiology of the upper airway in obstructive sleep apnea. Operative Techniques in Otolaryngology-Head and Neck Surgery, 2015; 26(2):74-77
- [Background] Wimms A, Woehrle H, Ketheeswaran S, Ramanan D, Armitstead J. Obstructive Sleep Apnea in Women: Specific Issues and Interventions. Biomed Res Int. 2016;2016:1764837. doi: 10.1155/2016/1764837. Epub 2016 Sep 6. PMID 27699167
- [Background] Senaratna CV, Perret JL, Lodge CJ, Lowe AJ, Campbell BE, Matheson MC, Hamilton GS, Dharmage SC. Prevalence of obstructive sleep apnea in the general population: A systematic review. Sleep Med Rev. 2017 Aug;34:70-81. doi: 10.1016/j.smrv.2016.07.002. Epub 2016 Jul 18. PMID 27568340
- [Background] Demir A, Ursavaş A, Aslan AT, Gülbay B, et al. Türk Toraks Derneği Obstrüktif Uyku Apne Sendromu Tanı Ve Tedavi Uzlaşı Raporu. Türk Toraks Dergisi 2012;13 EK 1 vol 13:5-9
- [Background] Lacasse Y, Godbout C, Series F. Health-related quality of life in obstructive sleep apnoea. Eur Respir J. 2002 Mar;19(3):499-503. doi: 10.1183/09031936.02.00216902. PMID 11936529
- [Background] Vanek J, Prasko J, Genzor S, Ociskova M, Kantor K, Holubova M, Slepecky M, Nesnidal V, Kolek A, Sova M. Obstructive sleep apnea, depression and cognitive impairment. Sleep Med. 2020 Aug;72:50-58. doi: 10.1016/j.sleep.2020.03.017. Epub 2020 Mar 23. PMID 32544796
- [Background] Bradley TD, Floras JS. Obstructive sleep apnoea and its cardiovascular consequences. Lancet. 2009 Jan 3;373(9657):82-93. doi: 10.1016/S0140-6736(08)61622-0. Epub 2008 Dec 26. PMID 19101028
- [Background] Gami AS, Howard DE, Olson EJ, Somers VK. Day-night pattern of sudden death in obstructive sleep apnea. N Engl J Med. 2005 Mar 24;352(12):1206-14. doi: 10.1056/NEJMoa041832. PMID 15788497
- [Background] Jordan AS, White DP, Owens RL, Eckert DJ, Rahangdale S, Yim-Yeh S, Malhotra A. The effect of increased genioglossus activity and end-expiratory lung volume on pharyngeal collapse. J Appl Physiol (1985). 2010 Aug;109(2):469-75. doi: 10.1152/japplphysiol.00373.2010. Epub 2010 May 27. PMID 20507968
- [Background] Iftikhar IH, Bittencourt L, Youngstedt SD, Ayas N, Cistulli P, Schwab R, Durkin MW, Magalang UJ. Comparative efficacy of CPAP, MADs, exercise-training, and dietary weight loss for sleep apnea: a network meta-analysis. Sleep Med. 2017 Feb;30:7-14. doi: 10.1016/j.sleep.2016.06.001. Epub 2016 Jun 28. PMID 28215266
- [Background] van Zeller M, Severo M, Santos AC, Drummond M. 5-years APAP adherence in OSA patients--do first impressions matter? Respir Med. 2013 Dec;107(12):2046-52. doi: 10.1016/j.rmed.2013.10.011. Epub 2013 Oct 16. PMID 24169074
- [Background] Donovan LM, Boeder S, Malhotra A, Patel SR. New developments in the use of positive airway pressure for obstructive sleep apnea. J Thorac Dis. 2015 Aug;7(8):1323-42. doi: 10.3978/j.issn.2072-1439.2015.07.30. PMID 26380760
- [Background] Geddes EL, O'Brien K, Reid WD, Brooks D, Crowe J. Inspiratory muscle training in adults with chronic obstructive pulmonary disease: an update of a systematic review. Respir Med. 2008 Dec;102(12):1715-29. doi: 10.1016/j.rmed.2008.07.005. Epub 2008 Aug 15. PMID 18708282
- [Background] Aslan GK, Gurses HN, Issever H, Kiyan E. Effects of respiratory muscle training on pulmonary functions in patients with slowly progressive neuromuscular disease: a randomized controlled trial. Clin Rehabil. 2014 Jun;28(6):573-81. doi: 10.1177/0269215513512215. Epub 2013 Nov 25. PMID 24275453
- [Background] Lin HC, Chiang LL, Ong JH, Tsai KL, Hung CH, Lin CY. The effects of threshold inspiratory muscle training in patients with obstructive sleep apnea: a randomized experimental study. Sleep Breath. 2020 Mar;24(1):201-209. doi: 10.1007/s11325-019-01862-y. Epub 2019 May 21. PMID 31115739
- [Background] Nobrega-Junior JCN, Dornelas de Andrade A, de Andrade EAM, Andrade MDA, Ribeiro ASV, Pedrosa RP, Ferreira APL, de Lima AMJ. Inspiratory Muscle Training in the Severity of Obstructive Sleep Apnea, Sleep Quality and Excessive Daytime Sleepiness: A Placebo-Controlled, Randomized Trial. Nat Sci Sleep. 2020 Dec 2;12:1105-1113. doi: 10.2147/NSS.S269360. eCollection 2020. PMID 33293881
- [Background] Erturk N, Calik-Kutukcu E, Arikan H, Savci S, Inal-Ince D, Caliskan H, Saglam M, Vardar-Yagli N, Firat H, Celik A, Yuce-Ege M, Ardic S. The effectiveness of oropharyngeal exercises compared to inspiratory muscle training in obstructive sleep apnea: A randomized controlled trial. Heart Lung. 2020 Nov-Dec;49(6):940-948. doi: 10.1016/j.hrtlng.2020.07.014. Epub 2020 Aug 13. PMID 32800391
- [Background] Puhan MA, Suarez A, Lo Cascio C, Zahn A, Heitz M, Braendli O. Didgeridoo playing as alternative treatment for obstructive sleep apnoea syndrome: randomised controlled trial. BMJ. 2006 Feb 4;332(7536):266-70. doi: 10.1136/bmj.38705.470590.55. Epub 2005 Dec 23. PMID 16377643
- [Background] Hsu B, Emperumal CP, Grbach VX, Padilla M, Enciso R. Effects of respiratory muscle therapy on obstructive sleep apnea: a systematic review and meta-analysis. J Clin Sleep Med. 2020 May 15;16(5):785-801. doi: 10.5664/jcsm.8318. Epub 2020 Feb 6. PMID 32026802
- [Background] Vitacca M, Paneroni M, Braghiroli A, Balbi B, Aliani M, Guido P, Fanfulla F, Pertosa M, Ceriana P, Zampogna E, Raccanelli R, Sarno N, Spanevello A, Maniscalco M, Malovini A, Ambrosino N. Exercise capacity and comorbidities in patients with obstructive sleep apnea. J Clin Sleep Med. 2020 Apr 15;16(4):531-538. doi: 10.5664/jcsm.8258. PMID 32003743
- [Background] Mendelson M, Bailly S, Marillier M, Flore P, Borel JC, Vivodtzev I, Doutreleau S, Verges S, Tamisier R, Pepin JL. Obstructive Sleep Apnea Syndrome, Objectively Measured Physical Activity and Exercise Training Interventions: A Systematic Review and Meta-Analysis. Front Neurol. 2018 Feb 22;9:73. doi: 10.3389/fneur.2018.00073. eCollection 2018. PMID 29520251
- [Background] Norman JF, Von Essen SG, Fuchs RH, McElligott M. Exercise training effect on obstructive sleep apnea syndrome. Sleep Res Online. 2000;3(3):121-9. PMID 11382910
- [Background] Lins-Filho OL, Pedrosa RP, Gomes JML, Dantas Moraes SL, Vasconcelos BCE, Lemos CAA, Pellizzer EP. Effect of exercise training on subjective parameters in patients with obstructive sleep apnea: a systematic review and meta-analysis. Sleep Med. 2020 May;69:1-7. doi: 10.1016/j.sleep.2019.12.022. Epub 2020 Jan 14. PMID 32045849